CLINICAL TRIAL: NCT01732042
Title: Retinal Venous Pressure (RVP) in Normals
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: USB-2011-326
Record Dates: First submitted 2012-10-24; First posted 2012-11-22 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: retinal venous pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Determinate the standard values of the retinal venous pressure in a cohort of healthy subjects.

DETAILED DESCRIPTION:
The retinal venous pressure (RVP) is an increasingly important dimension in the clinical assessment of retinal blood flow.

In literature only very few and also divergent data on the retinal venous pressure in healthy volunteers are described. A normal value study will provide us with an up-to-date database.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* eye diseases
* systemic diseases
* term medication (except contraceptives)
* pregnancy
* allergies to the ingredients Alcaine, Tropicamide and Phenylephrine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-11; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Retinal venous pressure | 1 hour
  Quantification of the retinal venous pressure as a standard value in a cohort of healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Josef Flammer, MD, Study Director — University of Basel, Dept. of Ophthalmology
Locations (1):
- University of Basel, Dept. of Ophthalmology, Basel, Switzerland